CLINICAL TRIAL: NCT05434156
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Intravenous Doses of ELE-101 in Healthy Adult Participants (Part 1) and Part 2, Open-Label Study to Evaluate a Range of Pharmacodynamic Effects of a Single Intravenous Dose of ELE-101 in Patients With Major Depressive Disorder.
Brief Title: ELE-101 Safety & Tolerability Study in Healthy Participants and Patients With Depression
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eleusis Therapeutics (Industry)
Collaborators: Beckley Psytech Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ET1001-ELE-101; 2022-000150-29 (EudraCT Number)
Record Dates: First submitted 2022-06-15; First posted 2022-06-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteers; Major Depressive Disorder; Depression
Keywords: ELE-101; psilocin; ELE-Psilo; psilocybin; psychedelic
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Open label in Part 2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Part 1) (Experimental): A single 10-minute intravenous infusion of 0.25 mg ELE-101 or placebo (randomized as 6 active and 2 placebo)
  Interventions: Drug: ELE-101; Drug: ELE-101 Placebo
- Cohort 2 (Part 1) (Experimental): A single 10-minute intravenous infusion of 0.75 mg ELE-101 or placebo (randomized as 6 active and 2 placebo)
  Interventions: Drug: ELE-101; Drug: ELE-101 Placebo
- Cohort 3 (Part 1) (Experimental): A single 10-minute intravenous infusion of 2.0 mg ELE-101 or placebo (randomized as 6 active and 2 placebo)
  Interventions: Drug: ELE-101; Drug: ELE-101 Placebo
- Cohort 4 (Part 1) (Experimental): A single TBD minute intravenous infusion of TBD mg ELE-101 or placebo (randomized as 6 active and 2 placebo)
  Interventions: Drug: ELE-101; Drug: ELE-101 Placebo
- Cohort 5 (Part 1) (Experimental): A single TBD minute intravenous infusion of TBD mg ELE-101 or placebo (randomized as 6 active and 2 placebo)
  Interventions: Drug: ELE-101; Drug: ELE-101 Placebo
- Cohort 6 (Part 2) (Experimental): A single TBD minute intravenous infusion of TBD mg ELE-101
  Interventions: Drug: ELE-101

INTERVENTIONS:
Drug: ELE-101 — ELE-101 solution for intravenous infusion
Drug: ELE-101 Placebo — ELE-101 placebo matching solution for intravenous infusion
  Arms: Cohort 1 (Part 1); Cohort 2 (Part 1); Cohort 3 (Part 1); Cohort 4 (Part 1); Cohort 5 (Part 1)

SUMMARY:
A study to assess the safety and tolerability of a drug called ELE-101 and see how the body absorbs and removes the drug and how it affects the body in healthy adult participants (Part 1) and in patients with depression (Part 2).

DETAILED DESCRIPTION:
This is a 2-part study. Part 1 is a phase I, double-blind, placebo-controlled, randomized study to assess the safety, tolerability, pharmacokinetic (PK) profile, pharmacodynamic (PD) and subjective drug intensity (SDI) of single ascending intravenous (IV) doses of ELE-101 in healthy male and female adult participants. Part 2 is a Phase IIa, open-label study to evaluate a range of pharmacodynamic effects of a single intravenous dose of ELE-101 in patients with depression.

Healthy participants will receive either ELE-101 or placebo as an IV infusion in Part 1 and patients with MDD will receive ELE-101 as an IV infusion in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants aged 18 to 65 years, inclusive.
* Participants have a body mass index (BMI) of 18 to 35 kg/m2, inclusive.
* Participants are able and willing to give written informed consent, adhere to the compliance terms during participation in the study, undergo the examinations and testing set forth in the study Protocol and clearly and reliably communicate their subjective symptoms to the Investigator.
* Part 2 Only: Patient has a diagnosis of MDD and is not on antidepressant medication.

Exclusion Criteria:

* Current, or history (within the last 6 months) of, alcohol or substance use disorder.
* Use of pharmacological compounds for psychiatric or neurological conditions acting on the CNS within 30 days or 5 half-lives (whichever is longer) prior to Screening.
* Current or clinically relevant history of schizophrenia, psychotic, bipolar disorder, delusional disorder, paranoid personality disorder, schizoaffective disorder, borderline personality disorder or panic disorder.
* In first-degree relatives, a history of schizophrenia, psychosis, bipolar disorder, delusional disorder, paranoid personality disorder or schizoaffective disorder.
* History of a diagnosis of Hallucinogen Persistent Perceptual Disorder (HPPD).
* Significant suicide risk.
* Other personal circumstances and behavior that is incompatible with establishment of rapport or safe exposure to psilocin, as judged by the Investigator.
* Part 1 Only: Ongoing current MDD, or history of MDD within the last year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Part 1: Percentage of participants with at least one safety event | Baseline up to Day 8
  * Safety will be evaluated by the monitoring of adverse events (AEs), vital signs, blood pressure, heart rate, pulse oximetry, electrocardiogram (ECG) evaluations, clinical laboratory assessments, injection site reactions and physical examination findings.
  * Suicidal ideation and behavior will be evaluated using the Columbia-Suicide Severity Rating Scale (C-SSRS).
  * Percentage of participants who experience at least one treatment-emergent adverse event (TEAE) will be captured.
  * Tolerability will be measured using the SDI questionnaires to rate the intensity of the psychedelic experience alongside recordings of anticipated adverse effects such as nausea and headache.
Part 2: Subjective Drug Intensity Ratings | pre-dose and at multiple time-points up to 24 hours post-dose
  - The SDI questionnaire will be used to rate the real-time intensity of the psychedelic experience

SECONDARY OUTCOMES:
Part 1 and 2: Cmax: Maximum observed plasma concentration for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: Tmax: Time to reach maximum plasma concentration (Cmax) for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: AUCinf: Area under the plasma concentration-time curve from Time 0 to Infinity for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: AUClast: Area under the plasma concentration-time curve from Time 0 to the time of the last quantifiable concentration for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: AUC0-24: Area under the plasma concentration-time curve from Time 0 to 24 hours for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: VZ: volume of distribution during the terminal disposition phase for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: VZss: volume of distribution at steady state for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: Cl: apparent total clearance from plasma for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: MRTinf: mean residence time from Time 0 to Infinity for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: t1/2: Terminal disposition phase half-life for ELE-101 and its metabolites | pre-dose and at multiple time-points up to 24 hours post-dose
  PK parameters in plasma will be calculated for psilocin and its primary metabolites throughout the study
Part 1 and 2: Dischargeability: Assessment of subject-discharge readiness | post-dose and 24 hours post-dose
  The dischargeability evaluation will be based on Investigator judgement after review of participant safety data.
Part 1: The dose related psychoactive effects of ELE-101 as evaluated by a Visual Analogue Scale | pre-dose and at multiple time-points up to 24 hours post-dose
  The Subjective Drug Intensity (SDI) is a Visual Analogue Scale scored from 0-10.
Part 2: The effects of ELE-101 on the severity of depression evaluated by the Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline up to Day 85
  The MADRS is a diagnostic questionnaire with ten items for measuring the severity of depressive episodes in patients with mood disorders. A higher MADRS score indicates more severe depression, and each item is scored from 0 to 6. The overall score ranges from 0 to 60.
Part 2: Percentage of participants with at least one safety event | Baseline up to Day 85
  * Safety will be evaluated by the monitoring of adverse events (AEs), vital signs, blood pressure, heart rate, pulse oximetry, electrocardiogram (ECG) evaluations, clinical laboratory assessments, injection site reactions and physical examination findings.
  * Suicidal ideation and behavior will be evaluated using the Columbia-Suicide Severity Rating Scale (C-SSRS).
  * Percentage of participants who experience at least one treatment-emergent adverse event (TEAE) will be captured.
  * Tolerability will be measured using the SDI questionnaires to rate the intensity of the psychedelic experience alongside recordings of anticipated adverse effects such as nausea and headache.

CONTACTS AND LOCATIONS:
Overall Officials: Neel Bhatt, Principal Investigator — MAC Clinical Research
Locations (2):
- United Kingdom (2):
  - MAC Clinical Research, Liverpool
  - MAC Clinical Research, Manchester

IPD SHARING:
Plan to Share IPD: No